CLINICAL TRIAL: NCT02815735
Title: Multi-Centre Clinical Evaluation of Two Reusable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-68 (VISA-407)
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A (Experimental): Participants wear comfilcon A lens for 4 weeks during the cross over study.
  Interventions: Device: comfilcon A
- lotrafilcon B (Active Comparator): Participants wear lotrafilcon B lens for 4 weeks during the cross over study.
  Interventions: Device: lotrafilcon B

INTERVENTIONS:
Device: comfilcon A — contact lens
  Arms: comfilcon A
Device: lotrafilcon B — contact lens
  Arms: lotrafilcon B

SUMMARY:
The aim of this study is to compare the subjective performance of the comfilcon A contact lens against lotrafilcon B contact lens after 4 weeks of reusable lens wear.

DETAILED DESCRIPTION:
This will be a 80 subject, randomized, bilateral, double-masked, dispensing, cross-over study comparing comfilcon A versus lotrafilcon B lenses over 4 weeks of daily wear for each lens pair.

ELIGIBILITY:
Inclusion Criteria:

* Spherical distance CL (Contact Lens) prescription between -1.00 and -6.00D (Diopter) OR in both eyes (inclusive)
* Adapted soft CL wearers (i.e. >1 month) who are reusable lens wearers*
* Spectacle cylinder 0.75D in both eyes
* Correctable to 6/9 in both eyes
* Be between 18 and 34 years of age (inclusive)
* Able to read, comprehend and sign an informed consent
* Own a mobile phone and be able to respond to SMS survey during the period 8am - 8pm
* Willing to comply with the wear and study visit schedule

Exclusion Criteria:

Any of the following will render a subject ineligible for inclusion:

* Existing wearer of daily disposable contact lenses
* Known allergy to Opti-Free PureMoist multipurpose solution
* Any active corneal infection, injury or inflammation
* Systemic or ocular allergies, which might interfere with CL wear
* Systemic disease, which might interfere with CL wear
* Ocular disease, which might interfere with CL wear
* Strabismus or amblyopia
* Subjects who have undergone corneal refractive surgery
* Subjects with keratoconus or other severe corneal irregularity contraindicating lens wear
* Pregnant, planning a pregnancy or lactating
* Use of systemic/topical medication contraindicating CL wear
* Diabetic
* Site employees or family members of investigators
* Participation in any concurrent trial or in the last 30 days

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Study Director — Visioncare Research Ltd.
Locations (9):
- United Kingdom (9):
  - Eyesite, Reading, Berkshire
  - Brock and Houlford, Chew Magna, Bristol
  - Tempany's Boutique Opticians, Broadstone, Dorset
  - Chalmers Opticians, Cardiff, Glamorgan
  - Leightons, St Albans, Hertfordshire
  - David Gould Opticians, Rawtenstall, Lancashire
  - Harrold Opticians, Uxbridge, Middlesex
  - Boots Opticians Ltd, Birmingham, Warwickshire
  - Visioncare Research Ltd., Farnham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects were not dispensed lenses due to screen failure. Seven subjects discontinued from the study due to the investigational site withdrawing from the study.
Groups:
- Comfilcon A, Then Lotrafilcon B: Participants wear comfilcon A lens, then lotrafilcon B for 4 weeks during the cross over study.
  comfilcon A: contact lens
  lotrafilcon B: contact lens
- Lotrafilcon B, Then Comfilcon A: Participants wear lotrafilcon B lens, then comfilcon A lens for 4 weeks during the cross over study.
  lotrafilcon B: contact lens
  comfilcon A: contact lens
Period: First Intervention (4 Weeks)
Arm/Group | Comfilcon A, Then Lotrafilcon B | Lotrafilcon B, Then Comfilcon A
Started | 36 | 38
Completed | 34 | 37
Not Completed | 2 | 1
Not completed — Discomfort | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Poor fitting characteristics | 0 | 1
Period: Second Intervention (4 Weeks)
Arm/Group | Comfilcon A, Then Lotrafilcon B | Lotrafilcon B, Then Comfilcon A
Started | 34 | 37
Completed | 33 | 37
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Participants wear comfilcon A and lotrafilcon B lens for 4 weeks during the cross over study.
  comfilcon A: contact lens
  lotrafilcon B: contact lens
Arm/Group | Overall Participants
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Comfort (insertion, end of the day, and overall) for habitual lenses assessed at baseline and comfilcon A and lotrafilcon B lenses assessed at 2 weeks and 4 weeks. Scale 0-10, 0=painful, 10=can't feel the lenses.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual (Baseline): Habitual data assessed at baseline.
- Comfilcon A (2 Weeks); Comfilcon A (4 Weeks): Participants wear comfilcon A lens for 4 weeks during the cross over study.
  comfilcon A: contact lens
- Lotrafilcon B (2 Weeks); Lotrafilcon B (4 Weeks): Participants wear lotrafilcon B lens for 4 weeks during the cross over study.
  lotrafilcon B: contact lens
Arm/Group | Habitual (Baseline) | Comfilcon A (2 Weeks) | Lotrafilcon B (2 Weeks) | Comfilcon A (4 Weeks) | Lotrafilcon B (4 Weeks)
Number analyzed (Participants) | 73 | 71 | 69 | 70 | 70
units on a scale
  Comfort on insertion | 8.90 (1.38) | 9.03 (1.10) | 8.70 (1.57) | 8.74 (1.25) | 8.60 (1.62)
  Overall comfort | 8.86 (1.38) | 8.13 (1.69) | 8.43 (1.54) | 8.11 (1.57) | 8.24 (1.65)
  End-of-Day Comfort | 8.03 (1.78) | 7.31 (2.21) | 7.45 (2.23) | 7.23 (2.17) | 7.34 (2.34)

2. Primary Outcome: Comfort During the Day
Description: Comfort during the day for comfilcon A and lotrafilcon B lenses assessed via via SMS (short message service) text message at days 3,12, and 26 at hours 8:00 am, 12:00 pm, 4:00 pm, and 8:00 pm. Scale 0-10, 0=painful, 10=can't feel the lenses.
Time Frame: Days 3, 12, 26
Population: Missing data from one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A (Day 3); Comfilcon A (Day 12); Comfilcon A (Day 26): Participants wear comfilcon A lens for 4 weeks during the cross over study.
  comfilcon A: contact lens
- Lotrafilcon B (Day 3); Lotrafilcon B (Day 12); Lotrafilcon B (Day 26): Participants wear lotrafilcon B lens for 4 weeks during the cross over study.
  lotrafilcon B: contact lens
Arm/Group | Comfilcon A (Day 3) | Lotrafilcon B (Day 3) | Comfilcon A (Day 12) | Lotrafilcon B (Day 12) | Comfilcon A (Day 26) | Lotrafilcon B (Day 26)
Number analyzed (Participants) | 69 | 69 | 72 | 70 | 70 | 68
units on a scale
  8:00 am | 8.98 (1.34) | 8.78 (1.60) | 8.67 (1.21) | 8.96 (1.26) | 8.78 (1.00) | 8.59 (1.48)
  12:00 pm | 8.94 (1.48) | 8.95 (1.22) | 8.59 (1.26) | 8.73 (1.41) | 8.72 (1.39) | 8.60 (1.32)
  4:00 pm: number analyzed (Participants) | 68 | 68 | 72 | 70 | 70 | 68
  4:00 pm | 8.51 (1.58) | 8.74 (1.31) | 8.51 (1.49) | 8.70 (1.45) | 8.31 (1.56) | 8.27 (1.62)
  8:00 pm: number analyzed (Participants) | 68 | 68 | 72 | 70 | 70 | 68
  8:00 pm | 8.15 (1.94) | 8.14 (1.59) | 7.91 (1.89) | 8.25 (1.77) | 7.85 (1.70) | 7.89 (1.92)

ADVERSE EVENTS:
Arm/Group | Comfilcon A | Lotrafilcon B
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other